CLINICAL TRIAL: NCT04529707
Title: Sleep Health Dysfunction and the Use of a Transdiagnostic Sleep Intervention in Duchenne Muscular Dystrophy
Brief Title: Sleep Intervention in Young Boys with Duchenne Muscular Dystrophy
Acronym: DMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Angela Caldwell, Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20030019
Record Dates: First submitted 2020-08-17; First posted 2020-08-28 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; Sleep; Intervention
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Intervention Model Description: The overall objective of this project is to conduct an early phase single-group repeated measures design project examining the implementation and within-subjects effects of a 10-week parent-mediated TranS-CY program to improve sleep health in young boys with DMD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sleep Intervention (Experimental): All participants will engage in a 10-week, parent mediated sleep intervention with weekly education sessions.
  Interventions: Behavioral: Transdiagnostic Behavioral Sleep Intervention

INTERVENTIONS:
Behavioral: Transdiagnostic Behavioral Sleep Intervention — The Transdiagnostic Sleep and Circadian Intervention for Youth (TranS-CY) uses a comprehensive sleep health framework along with robust evidence for promoting healthy sleep patterns in youth. The TranS-CY incorporates best practices from numerous efficacious behavioral sleep interventions including 1) cognitive behavioral therapy, 2) interpersonal and social rhythm therapy, and 3) behavioral treatment of circadian rhythm sleep-wake disorders. The "traditional" TranS-CY is clinician-led and provides a robust sleep treatment framework for youth with a wide range of disorders and sleep health concerns. For this study, investigators are using the basic framework of the TranS-CY, but clinicians will train parents to incorporate the intervention into the home for their young child with DMD. Trained clinicians will work with parents to ensure the basic components of the TranS-CY are incorporated into the home-based intervention.

SUMMARY:
This project will systematically plan and evaluate the implementation of the Transdiagnostic Sleep and Circadian Intervention for youth (TranS-CY). As an early stage study, investigators will focus on recruitment strategies to reach the target population and collection of preliminary data on primary and secondary effects of the TranS-CY. Weekly remote (video web conferencing) parent training sessions will allow investigators to explore adoption through parent adherence and examine whether the essential elements of the TranS-CY intervention (e.g., motivational interviewing, goal setting, problem solving, sleep routine scheduling, monitoring) can be consistently taught by clinicians and implemented by parents into the home setting.

DETAILED DESCRIPTION:
Pre-phase (2 weeks in duration):

Initial Interview: Following informed consent and enrollment, participants will complete a 45-60 minute interview with research investigators using video web conferencing (e.g., Zoom). If the participant agrees, this interview will be recorded. During this interview, investigators will gather descriptive data to characterize the sample including information regarding: 1) the child (age, disease severity for DMD, weight/ height, race/ethnicity, location (rural/suburban/urban), grade in school, medication use); 2) the parent (race/ethnicity, marital status, work status, education level, income); 3) the child's sleep environment (technology/telephone access, darkness, temperature, bed/bedroom sharing); 4) the child's daily activities and routines (current wake-up time & routines; activities in the home; activities at school and after school); and 5) the child's nighttime routines (activities prior to bedtime; current bedtime routine; technology use prior to bedtime).

ActiGraph: Each parent-child dyad will be mailed a package containing the Actigraph GT9x with wristband, charging device, a manual of operating procedures (MOP) providing all technical and protocol instructions, and phone numbers for research team support. Throughout the 2-week pre-phase data collection period, parents will be required to log and push data from their child's Actigraph to a secure cloud service, CentrePoint, via Wi-Fi each day. This will be accomplished through an app and all data will be de-identified.

Intervention Implementation Phase (10-week duration):

Training Modules: During the intervention phase, weekly video-conference meetings will be held where trained clinicians will guide parents through approximately 60-minute web-based modules using a video-conferencing platform (e.g., Zoom). These sessions will focus on education, dynamic parent training (child-related goal-setting and problem-solving), assessment of sleep health dimensions, and development of a weekly sleep and activity diary. Parents will be provided with a personalized TranS-CY Parent Workbook, which contains information regarding each of the 10 weekly modules. Each weekly session will be agenda driven with the option to revise the agenda based on family needs. Children/youth with DMD will be invited to attend the sessions and provide as much feedback as possible. Data will be collected on parent attendance to assess intervention adoption. Each week, clinicians will request feedback on the previous week's session and provide additional educational support for the previous content should it be required.

Intervention Questionnaires: During the 10-week intervention phase, parents will be asked to complete knowledge checks every 2-3 weeks in order to confirm understanding of the module information (primary outcome). These questionnaires will either be asked verbally during the session or questions will be sent to the parent's email through Qualtrics, a HIPAA compliant survey software platform. Hard copies of the knowledge checks will be sent if the parent prefers.

Sleep and Activity Log: Throughout the intervention phase, parents will be asked to complete a daily sleep and activity log covering their child's day. This log will be sent to their emails using Qualtrics. Each log will take approximately 3-5 minutes to complete.

Post-Intervention Phase (2 weeks):

ActiGraph: At the end of the 10-week intervention, each participant (parent-child dyad) will again be mailed an Actigraph GT9x, all accessories and protocols. Throughout the 2-week post-phase data collection period, parents will again use their personal smart-phone app to log and push data from the Actigraph to CentrePoint, via Wi-Fi each day. Data from the Actigraph GT9x will be provide the secondary outcome of percent sleep efficiency. Investigators will explore change in percent sleep efficiency at pre-post 10 week TranS-CY intervention.

ELIGIBILITY:
Inclusion Criteria:

* Parents/caregivers of youth between ages 6 and 17 with a primary diagnosis of Duchenne muscular dystrophy (DMD) who lives at home .
* Access to a smart-phone or computer and internet for the weekly web-based sessions, as well as uploading of the Actigraph data;
* English speaking.

Exclusion Criteria:

* Unable to speak or read English
* Their child with DMD has cognitive or behavioral concerns that would limit participation and follow-through of intervention;
* Their child/youth with DMD is currently receiving an intervention for a sleep related disorder

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Parent Mastery Questionnaire | A 10-item questionnaire focused on intervention modules will be delivered every 2-3 weeks during the 10 week intervention. Parents will be required to answer questions that address their knowledge of the information provided in each module.
  100% of parents who are retained throughout the study will attain ≥80% knowledge accuracy at each knowledge check time point and will accurately answer 8 of the 10 questions provided.

SECONDARY OUTCOMES:
Child intradaily variability from Actigraphy | 2 weeks pre-intervention and 2 weeks post-intervention
  Vector magnitude scores from Actigraphy for each 2-week data collection period (pre and post intervention) are analyzed through nParAct software. Analyses provide us with our secondary outcome of intradaily variability. Intradaily variability is the frequency and extent of transitions between periods of rest and activity on an hourly basis over 24 hours. Relative amplitude is how active a child is during a 24 hour period.
Child relative amplitude from Actigraph | 2 weeks pre-intervention and 2 weeks post-intervention.
  Vector magnitude scores from Actigraphy for each 2-week data collection period (pre and post intervention) are analyzed through nParAct software. Analyses provide us with our secondary outcome of relative amplitude. Relative amplitude is how active a child is during a 24 hour period.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Caldwell, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
This is a preliminary study focused on determining if the TranS-CY can be modified and implemented into the home by parents of young boys with DMD. The primary and secondary outcomes are focused on collecting data regarding parent knowledge of the intervention components and change in intradaily variability and relative amplitude (through Actigraphy) of the child with DMD pre and post intervention.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and additional supporting information will be made available approximately 3 months after summary data are published or otherwise disseminated.
Access Criteria: IPD will be shared with researchers within and outside of the University of Pittsburgh through email requests to the lead principal investigator. The University of Pittsburgh may require a data use agreement be developed and signed by both institutions. The full study protocol and informed consent forms will be shared. Only aggregate and de-identified data collected throughout the clinical trial will be shared.